CLINICAL TRIAL: NCT00856453
Title: Restorative Yoga for Women With Ovarian Cancer Undergoing Chemotherapy
Brief Title: Yoga in Relieving Fatigue in Patients Undergoing Chemotherapy for Ovarian Cancer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: slow accrual
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CDR0000632845; CCCWFU-98408; IRB00007745
Record Dates: First submitted 2009-03-04; First posted 2009-03-05 (Estimated); Last update posted 2018-08-09 (Actual); Status verified 2018-08

CONDITIONS: Depression; Fatigue; Ovarian Cancer
Keywords: fatigue; depression; recurrent ovarian epithelial cancer; recurrent ovarian germ cell tumor; stage I ovarian epithelial cancer; stage I ovarian germ cell tumor; stage II ovarian epithelial cancer; stage II ovarian germ cell tumor; stage III ovarian epithelial cancer; stage III ovarian germ cell tumor; stage IV ovarian epithelial cancer; stage IV ovarian germ cell tumor
MeSH Terms: conditions — Depression; Fatigue; Ovarian Neoplasms; Carcinoma, Ovarian Epithelial

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Yoga classes plus home yoga practic (Experimental)
  Interventions: Behavioral: Home yoga practice; Behavioral: yoga classes
- home yoga practice alone (Experimental)
  Interventions: Behavioral: Home yoga practice

INTERVENTIONS:
Behavioral: Home yoga practice — training for and tracking of patient's practice of yoga at home
Behavioral: yoga classes — organized out of home classes for yoga
  Arms: Yoga classes plus home yoga practic

SUMMARY:
RATIONALE: Yoga may decrease fatigue, distress, and depression, and improve sleep quality in patients undergoing chemotherapy for ovarian cancer. It is not yet known whether practicing yoga in group classes is more effective than practicing yoga at home.

PURPOSE: This randomized clinical trial is studying how well yoga works in relieving fatigue in patients undergoing chemotherapy for ovarian cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Examine the effectiveness of a restorative yoga (RY) intervention vs home yoga practice in patients undergoing chemotherapy for ovarian cancer.

Secondary

* Examine the effectiveness of RY vs home yoga practice on depression, distress, and sleep quality in these patients.
* Examine the acute (pre- and post-yoga class) effects in these patients.
* Test the feasibility of using behavioral strategies to enhance yoga intervention adherence.

OUTLINE: Patients are randomized to 1 of 2 arms.

* Arm I (restorative yoga intervention): Patients attend 45-minute group yoga classes every 3 weeks on the days they are scheduled for chemotherapy for approximately 5-6 sessions. Patients are provided with a yoga DVD, a manual with photos and written descriptions/guidance to practice yoga postures at home, and basic yoga equipment (yoga mat, strap, block, yoga blankets) and instructed to practice to the DVD 3 times per week (twice weekly during week of group yoga class) for ≥ 45 minutes. Patients record yoga practice time/activity at the third yoga session of each week.
* Arm II (home yoga practice): Patients are provided with a yoga DVD, a manual with photos and written descriptions/guidance to practice yoga postures at home, and basic yoga equipment (yoga mat, strap, block, yoga blankets) and instructed to practice to the DVD 3 times per week for ≥ 45 minutes. Patients record yoga practice time/activity at the third yoga session of each week.

All patients complete questionnaires at baseline, at weeks 9, 18, and 22. Self-report measures include Distress Thermometer, Positive and Negative Affect Schedule, Center for Epidemiologic Studies-Depression Scale, M.D. Anderson Symptom Inventory, Functional Assessment of Cancer Therapy - Ovarian, Functional Assessment of Chronic Illness Therapy (FACIT) - Spiritual Subscale, FACIT- Fatigue Subscale, State-Trait Anxiety Inventory, Women's Health Initiative Insomnia Rating Scale, Medical Outcome Study-Social Support Survey, Integrative Medicine Use, Pre- and Post- Class Ratings, and Intervention Feedback .

After completion of study, patients are followed at 4 weeks.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of ovarian cancer

  * Any stage disease
* Must be between 2-24 months post-primary treatment (surgery) following initial diagnosis and/or have a recurrence of ovarian cancer within the past 24 months (irrespective of current treatment status)
* Began a new chemotherapy treatment regimen within the past 4 weeks or planning to begin new chemotherapy treatment regimen within the next 4 weeks

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Physically able to attend the intervention classes
* Able to understand written and spoken English
* Agree to keep psychiatric medications and doses stable during study intervention
* No medical contraindications reported by the attending physician
* No bipolar disorder, schizophrenia, psychotic depression, or any other psychotic disorder
* No usage of illicit drugs

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* More than 3 months since prior yoga practice

Ages: 18 Years to 120 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2009-05; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Self-reported fatigue | 22 weeks

SECONDARY OUTCOMES:
Self-reported distress, depression, and sleep quality | 22 weeks
Pre- and post-yoga class change in symptom/distress ratings | 22 weeks
Yoga intervention adherence | 18 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne C. Danhauer, PhD, Principal Investigator — Wake Forest University Health Sciences; Brigitte E. Miller, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Comprehensive Cancer Center, Winston-Salem, North Carolina, United States